# **Statistical Analysis Plan (SAP)**

**Study ID:** 213299

**Official Title of Study:** A Global, Molecular Disease Characterization Initiative (MDCI) in Oncology Clinical Trials

**Date of Document:** 29 Nov 2022

NCT number: NCT04772053

### **CONFIDENTIAL**

The GlaxoSmithKline group of companies

**Information Type:** Statistical Analysis Plan (SAP)



213299

### TITLE PAGE

**Protocol Title:** A Global, Molecular Disease Characterization Initiative

(MDCI) in Oncology Clinical Trials

**Study Number:** 213299

**Compound Number:** No Compound

**Abbreviated Title:** Molecular Disease Characterization Initiative (MDCI)

Sponsor Name: GSK Research & Development Limited

**Regulatory Agency Identifier Number(s)** 

**Registry** ID

Clintrials.gov NCT04772053

Copyright 2022 the GSK group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | INTR | ODUCTIO | ON | 4 |
| | 1.1. | | ves, Estimands and Endpoints | |
| | | 1.1.1. | Objectives and Endpoints | |
| | 1.2. | Study [ | Design | |
| 2. | STAT | ISTICAL | HYPOTHESES | 7 |
| | 2.1. | | city Adjustment | |
| 3. | ANAL | YSIS SE | TS | 7 |
| 4. | STAT | ISTICAL | ANALYSES | 7 |
| | 4.1. | | | |
| | | 4.1.1. | General Methodology | |
| | | 4.1.2. | Baseline Definition | |
| | 4.2 | | y Endpoint(s) Analyses | |
| | | | Definition of endpoint | |
| | | 4.2.2. | | |
| | 4.3. | | dary Endpoint(s) Analyses | |
| | CCI | | | |
| | 4.5. | Safety | Analyses | 8 |
| | | 4.5.1. | | |
| | | 4.5.2. | Adverse Events/Serious Adverse Events | 9 |
| | 4.6. | Interim | Analyses | |
| | 4.7. | Change | es to Protocol Defined Analyses | 9 |
| 5. | SAMI | PLE SIZE | DETERMINATION | 9 |
| 6. | SUPF | PORTING | DOCUMENTATION | 10 |
| | 6.1. Appendix 1 Study Population Analyses | | | |
| | | 6.1.1. | Participant Disposition | 10 |
| | | 6.1.2. | Demographic and Baseline Characteristics | 10 |
| | | 6.1.3. | Protocol Deviations | 10 |
| | 6.2. | Append | dix 2 Data Derivations Rule | 11 |
| | | 6.2.1. | Study Day and Reference Dates | 11 |
| | | 6.2.2. | Assessment Window | |
| | | 6.2.3. | Handling of Partial Dates | |
| | | 6.2.4. | Early PK Access Key Activities | |
| 7 | REE | DENCE | | 14 |

# **Version history**

| SAP<br>Version | Approval Date | Protocol<br>Version<br>(Date) on<br>which SAP<br>is Based | Change | Rationale |
|---|---|---|---|---|
| 1 | 29 Nov 2022 | Amendment<br>03 (25-Oct-<br>2021) | Not<br>Applicable | Original version |

## 1. INTRODUCTION

The purpose of this SAP is to describe the planned analyses to be included in the synoptic CSR and disclosure for Study 213299. Details of the planned analyses are provided.

## 1.1. Objectives, Estimands and Endpoints

Estimands are not applicable for this study.

## 1.1.1. Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary | |
| To evaluate molecular and immunological profile of tumor and peripheral blood of all enrolled participants, across indications and within tumor subsets (Building a GSK Clinical Science Database for tumor profiling and correlative studies). | Profile of patient specific selection biomarkers targeted by therapeutics with the GSK oncology pipeline, as well as other as detailed in the study reference manual (SRM). |
| CCI | |



## 1.2. Study Design



Footnotes: <sup>1</sup>MDCI will be an optional protocol under select GSK oncology protocols; <sup>2</sup>In the case that Visit 1 and 2 are combined, all corresponding samples must be collected per the SoA (Protocol Section 1.3) at this visit and after eligibility is confirmed; <sup>3</sup>Subset of data to be shared on Gather Share Know; <sup>4</sup>Patient's molecular profile and medical history will be compared against the eligibility criteria of select GSK oncology protocols to identify potential trial options; <sup>5</sup>Visit 3 may occur remotely via



| Overview of Study Design and Key Features | |
|---|---|
| Study | Not applicable |
| intervention | |
| Study | Not applicable |
| intervention | |
| Assignment | |
| Interim | Due to the continuous nature of this study, there is no interim analysis |
| Analysis | phase. |

### 2. STATISTICAL HYPOTHESES

MDCI is an study and a pre-screening protocol. The analysis will be descriptive in nature. No formal hypothesis testing is planned under this study.

## 2.1. Multiplicity Adjustment

No formal statistical testing will be performed; therefore, no adjustments for multiplicity are planned.

### 3. ANALYSIS SETS

| Analysis Set | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All participants who sign the ICF | <ul> <li>Study population</li> </ul> |
| Enrolled | All participants who sign the ICF and<br>meet inclusion/exclusion criteria | Study Population Safety |

### 4. STATISTICAL ANALYSES

#### 4.1. General Considerations

Unless and otherwise specified, only the study column will be reported in summary tables.

### 4.1.1. General Methodology

Unless otherwise specified, continuous data will be summarized using descriptive statistics: n, mean, standard deviation (std), median, minimum and maximum.

Categorical data will be summarized as the number and percentage of participants in each category.

It is anticipated that patient accrual will be spread thinly across centres and summaries of data by centre would unlikely be informative and will not, therefore, be provided.

### 4.1.2. Baseline Definition

No endpoints/summary measures are reported which requires baseline definition. Hence, not applicable.

## 4.2. Primary Endpoint(s) Analyses

### 4.2.1. Definition of endpoint

Profile of patient-specific selection biomarkers that are targeted by therapeutics within the GSK oncology pipeline, as well as other study reference manual (SRM).

### 4.2.2. Main analytical approach

"Enrolled" analysis set will be used to perform primary endpoint analysis.

A summary table containing biomarker status of participants will be provided. Biomarker status includes Inducible T-cell Co-Stimulator (ICOS) status, New York esophageal squamous cell carcinoma 1 (NY-ESO-1)/Cancer testis antigen 2 (LAGE-1a) status and Programmed death protein 1 Ligand (PD-L1) status.

This summary table contains number and percentage of participants with positive/negative status by biomarker (ICOS, NY-ESO-1/LAGE-1a and PD-L1).

A subject level listing containing biomarker status of participants will also be provided.

## 4.3. Secondary Endpoint(s) Analyses

Not applicable, as there are no secondary endpoints defined under this protocol.



## 4.5. Safety Analyses

The safety analyses will be based on the Enrolled Analysis Set, unless otherwise specified.

Only the AEs/SAEs related to study procedures are collected in this study. If there are no AEs/SAEs in the database, a standard 'No data to report' display will be generated.

### 4.5.1. Extent of Exposure

Not applicable.

#### 4.5.2. Adverse Events/Serious Adverse Events

Adverse events analyses including the analysis of adverse events (AEs), serious adverse events (SAEs) will be based on GSK Core Data Standards. Adverse events will be coded using the standard Medical Dictionary for Regulatory Affairs (MedDRA dictionary) and grouped by system organ class (SOC). Adverse events will be graded by the investigator according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v5.0).

An overview summary of AEs, including counts and percentages of participants with any AE will be created by SOC and PT.

All SAEs will be tabulated based on the number and percentage of participants who experienced the event by SOC and PT. The summary of all SAEs will be created by SOC and PT.

A summary of fatal SAEs will also be provided.

A Summary of Fatal AEs and Non-serious AEs by SOC and PT will also be provided.

A listing of all AEs collected will be provided. SAE flags are included in the listing of all AEs. Separate supportive listings with participant level details will be generated for

- Fatal SAEs
- Non-Fatal SAEs.

### 4.5.2.1. Additional Safety Assessments

Routine safety assessments (e.g., ECG and vital signs) were only collected during screening. Other than the collection of AE information, no further safety assessments were mandated in the protocol after screening was complete. Therefore, no additional safety information will be summarised for this study.

## 4.6. Interim Analyses

Due to the continuous nature of this study, there is no interim analysis phase. Data will be continuously monitored and analysed in real-time during the course of the study.

## 4.7. Changes to Protocol Defined Analyses

There were no changes or deviations to the originally planned statistical analysis specified in the protocol amendment 3 (Dated: 25-OCT-2021).

#### 5. SAMPLE SIZE DETERMINATION

Since MDCI does not aim to test any specific hypothesis or answer any particular question, there is no statistical requirement to reach a specific number of samples and patients.

### 6. SUPPORTING DOCUMENTATION

## 6.1. Appendix 1 Study Population Analyses

Unless otherwise specified, the study population analyses will be based on the Enrolled Analysis Set.

### 6.1.1. Participant Disposition

A summary of the number of participants in each of the participant level analysis set mentioned in Section 3 will be provided.

A summary of subject status and reason for study withdrawal will be provided. This display will show the number and percentage of subjects who withdrew from the study, including primary reasons for study withdrawal. The Enrolled Analysis set will be used.

A summary and listing of screening status and reasons for screen failure will be provided using the Screened Analysis Set. Per GSK reporting standards, participants who were rescreened will appear once in these displays according to their final status.

## 6.1.2. Demographic and Baseline Characteristics

The demographic characteristics including age, gender, ethnicity, weight at screening and race will be summarized with descriptive statistics. In addition, the following age categories will be summarized: 18-64, 65-84 and >=85 based on the Enrolled Analysis Set.

A listing of demographic characteristics and race will be provided.

#### 6.1.3. Protocol Deviations

Important protocol deviations will be summarized.

Protocol deviations will be tracked by the study team throughout the conduct of the study. These protocol deviations will be reviewed to identify those considered as important as follows:

- Data will be reviewed prior to freezing the database to ensure all important deviations (where possible without knowing the study intervention details) are captured and categorised in the protocol deviations dataset.
- o This dataset will be the basis for the summaries of important protocol deviations.

If there is no data to report a standard "no data to report" displays will be produced.

## 6.2. Appendix 2 Data Derivations Rule

### 6.2.1. Study Day and Reference Dates

The reference date is the study enrolment date and will be used to calculate study day

The study day is calculated as below:

- Assessment Date = Missing → Study Day = Missing
- Assessment Date < Reference Date → Study Day = Assessment Date Ref Date
- Assessment Data ≥ Reference Date → Study Day = Assessment Date Ref Date + 1

#### 6.2.2. Assessment Window

No Assessment window will be applied.

## 6.2.3. Handling of Partial Dates

The partial date imputation will follow ADaM conventions. The ADaM approach is to populate the numeric date variables with the imputed date and add a flag variable to the dataset that indicates the level of imputation.

The flag variable can contain the values: blank, 'D', 'M', 'Y'.

blank: indicates that no imputation was done

D='Day': indicates that the day portion of the date is imputed

M='Month': indicates that the month and day portions of the date are imputed

Y='Year': indicates that the entire date (year, month, and day) is imputed

Example of date variables:

XYZD - character date variable

XYZDT - numeric date variable

XYZDTFL - flag variable

Details on imputing partial dates for specific datasets are outlined below

| Element | Reporting Detail | |
|---|---|---|
| General | <ul> <li>Partial dates we displays.</li> <li>However, whe temporary var partial dates me specific analys.</li> <li>Imputed partial onset or duration.</li> </ul> | al dates will be displayed as captured in participant listing anys. Ever, where necessary, display macros may impute dates as orary variables for sorting data in listings only. In addition, all dates may be imputed for 'slotting' data to study phases or for fic analysis purposes as outlined below. Ited partial dates will not be used to derive study day, time to or duration (e.g., time to onset or duration of adverse events), psed time variables (e.g., time since diagnosis). |
| Adverse Events | Partial dates for following con Missing start day | tes for AE recorded in the CRF will be imputed using the conventions: |
| | Missing start day and month | If study enrollment date is missing, then set start date = January 1. Else if study enrollment date is not missing: |

| Element | Reporting Detail | |
|---|---|---|
| | Missing end day | A '28/29/30/31' will be used for the day (dependent on the month and year). |
| | Missing end day and month | No Imputation |
| | Completely missing | No imputation |
| | start/end date | |

# 6.2.4. Early PK Access Key Activities

Not applicable.

# 7. REFERENCES

None